



IRAS ID: 242462

## **Informed Consent Form**

## Assessing gut permeability using spectroscopy

Study title: Non-invasive transcutaneous spectroscopy for the assessment of gut permeability (GutPerm)

IRAS Project ID: 242462

| Pa | atient Trial ID Number: | |
|---|---|---|
| Na | ame of Principal Investigator: <u>Dr Alex Thompson</u> | |
| Na | ame of patient to whom this ICF applies: | |
| | Please | initial boxes |
| 1. | I confirm that I have read and understand the Patient Information Sheet "Assessing gut permeability using spectroscopy v4.0 31-May-2018" for the above study and have had the opportunity to ask questions about the study and understand what is involved. | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time, without giving any reason, without my medical care or other legal rights being affected, and I understand that data collected up to the point of my withdrawal may still be used. | |
| 3. | I agree to have a 'Spectroscopic gut permeability test' and understand that there is a small risk of nausea and other allergic reactions (including anaphylaxis) with this test. | |
| 4. | I understand that sections of any of my medical notes may be looked at by authorised individuals from Imperial College Healthcare NHS Trust, from Imperial College London, or from regulatory authorities where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | |
| 5. | I agree to allow information about me to be collected, analysed, reported and transferred to other approved collaborators within and outside the European Economic Area for healthcare and/or medical research purposes. I understand that my identity will remain anonymous. | |
| 6. | I wish to be contacted by e-mail with a summary of the research findings once the study is complete. Your e-mail address will not be used for any other purpose. | |
| | Contact e-mail: | |
| | If you do <u>NOT</u> wish to be contacted regarding the study results, please put a line through all of point 6 above, do <u>NOT</u> leave a contact e-mail address and do <u>NOT</u> initial the box as indicated – you can still participate in the main trial. | |
| 7. | I agree to take part in the study. | |

Please sign and date overleaf.





| Name of Subject | Signature | Date |
|-------------------------------|-----------|----------|
| Name of Person taking consent | Signature | <br>Date |

1 copy for subject; 1 copy for Principal Investigator; 1 copy to be kept with hospital notes